| | Statistical Analysis Plan Fir |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | Phase IIIb randomized, open, controlled, multicenter study to evaluate the immunogenicity and safety of the RTS,S/AS01 <sub>E</sub> candidate malaria vaccine, when administered as primary vaccination at 6, 7.5 and 9 months of age with or without coadministration of measles, rubella and yellow fever vaccines followed by an RTS,S/AS01 <sub>E</sub> booster vaccination 18 months post Dose 3, to children living in sub-Saharan Africa. |
| eTrack study number and | 200596 (MALARIA-073) |
| Abbreviated Title Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 09-Apr-2018 |
| Co-ordinating author: | (Statistician) |
| Reviewed by: | Clinical and Epidemiology Project Lead) PPD (Clinical Research and Development Lead) PPD (Lead statistician) |
| | (Lead statisticiali) |
| | (Statistician) |
| | (Lead statistical analyst) |
| | (Scientific writer) |
| | (Lead Scientific writer) |
| | (Regulatory Affail) |
| | (SEKW physician) |
| | (SERIVI SCIERUSI) |
| Approved by | (Fublic disclosure Fivi) |
| Approved by: | (Clinical and Epidemiology Project Lead) delegating to PPD (Clinical Research and Development Lead) PPD (Lead statistician) |
| | (Lead Scientific writer) |
| | (Lead statistical analyst) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

200596 (MALARIA-073) Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | BBREVIATIONS | 10 |
| 1. | DOCU | JMENT HISTORY | 12 |
| 2. | STUD | Y DESIGN | 13 |
| 3. | OR IE | CTIVES | 17 |
| ٥. | 3.1. | Primary objective | |
| | 3.2. | | |
| | 3.3. | Tertiary objective | |
| 4. | | OINTS | 18 |
| | 4.1. | Primary endpoints | 18 |
| | 4.2. | Secondary endpoints | |
| | 4.3. | Tertiary endpoints | 21 |
| 5. | ANAL` | YSIS SETS | 22 |
| | 5.1. | Definition | 22 |
| | | 5.1.1. Enrolled Set | |
| | | 5.1.2. Exposed Set (ES) | 22 |
| | | 5.1.3. Per-Protocol Set for analysis of immunogenicity (PPS for immunogenicity) | 22 |
| | 5.2. | Criteria for eliminating data from Analysis Sets | |
| | 5.2. | 5.2.1. Elimination from Exposed Set (ES) | |
| | | 5.2.2. Elimination from Per-protocol analysis Set (PPS) | |
| | | 5.2.2.1. Excluded subjects | |
| | 5.3. | Important protocol deviation not leading to elimination from per- | 20 |
| | 0.0. | protocol analysis set | 24 |
| 6. | STATI | ISTICAL ANALYSES | 24 |
| ٠. | 6.1. | Demography | |
| | | 6.1.1. Analysis of demographics/baseline characteristics planned | |
| | | in the protocol | 24 |
| | | 6.1.2. Additional considerations | 24 |
| | 6.2. | Exposure | 25 |
| | | 6.2.1. Analysis of exposure planned in the protocol | 25 |
| | | 6.2.2. Additional considerations | 25 |
| | 6.3. | Efficacy/Effectiveness | |
| | | 6.3.1. Analysis of efficacy planned in the protocol | |
| | | 6.3.2. Additional considerations | |
| | 6.4. | Immunogenicity | |
| | | 6.4.1. Analysis of immunogenicity planned in the protocol | |
| | | 6.4.2. Additional considerations | |
| | 6.5. | Analysis of safety | |
| | | 6.5.1. Analysis of safety planned in the protocol | |
| | | 6.5.2. Additional considerations | 29 |
| | | 6.5.2.1. Concomitant Medication and Concomitant | 30 |

200596 (MALARIA-073) Statistical Analysis Plan Final

| | | | Statistical / trial year | , i idii i iiidi |
|---|---|---|---|---|
| 7. | ANAL | YSIS INTI | ERPRETATION | 30 |
| 8. | CONE | OUCT OF | ANALYSES | 31 |
| | 8.1. | Segueno | ce of analyses | 31 |
| | 8.2. | | al considerations for interim analyses | |
| 9. | CHAN | IGES FRO | OM PLANNED ANALYSES | 31 |
| 10. | LIST | OF FINAL | REPORT TABLES, LISTINGS AND FIGURES | 32 |
| 11. | ANNE | X 1 STAN | NDARD DATA DERIVATION RULE AND STATISTICAL | |
| | METH | IODS | | 33 |
| | 11.1. | Statistica | al Method References | |
| | | | Other references | |
| | 11.2. | | d data derivation | |
| | | | Date derivation | |
| | | | Dose number | |
| | | | Demography | |
| | | 11.2.4. | | |
| | | 11.2.5. | | |
| 12 | ANNE | X 2· SUM | IMARY ON ELIMINATION CODES | 39 |
| . 2. | , u 41 4L | ., . Z. OOW | With the Control of t | |
| 13 | ANNE | X 3· STU | DY SPECIFIC MOCK TFL | 41 |

200596 (MALARIA-073) Statistical Analysis Plan Final

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups and epochs foreseen in the study | 14 |
| Table 2 | Study groups and treatment foreseen in the study | 14 |
| Table 3 | Blinding of study epoch | 14 |
| Table 4 | Immunological read-outs | 15 |
| Table 5 | Reporting periods for adverse events and serious adverse events | 16 |
| Table 6 | Safety Sets | 39 |
| Table 7 | Immunogenicity Sets | 39 |

200596 (MALARIA-073) Statistical Analysis Plan Final

# **LIST OF FIGURES**

| | | PAGE |
|----------|--------------|------|
| Figure 1 | Study design | 13 |

200596 (MALARIA-073) Statistical Analysis Plan Final

# **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Number of subjects enrolled by center, per study group (Exposed Set) | 41 |
| Template 2 | Number of enrolled subjects by country (All Enrolled Set) | 41 |
| Template 3 | Number of enrolled subjects by age category (All Enrolled Set) | 41 |
| Template 4 | Consort, per study group (Month 4.5)(all screened set) | 42 |
| Template 5 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal until Month 4.5, per study group (Exposed Set) | 42 |
| Template 6 | Deviations from specifications for age and intervals between study visits (Exposed Set) | 43 |
| Template 7 | Number of subjects at each visit and list of withdrawn subjects until Month 4.5, per study group (Exposed Set) | 44 |
| Template 8 | Number and percentage of subjects who received study vaccine doses by vaccine, per study group (Exposed Set) | 45 |
| Template 9 | Number of subjects enrolled into the study as well as the number excluded from PPS analyses with reasons for exclusion, per study group (all enrolled set) | 46 |
| Template 10 | Summary of demographic characteristics at baseline, per study group (Exposed Set) | 47 |
| Template 11 | Minimum and maximum activity dates, per study group (Exposed Set) | 47 |
| Template 12 | Eligibility (Total cohort) (all screened set) | 48 |
| Template 13 | Primary objective assessment: Non-inferiority assessment of anti-CS antibody response to RTS,S/AS01E in Coad and RTS,S groups, GMT ratio, Month 4 (Per-Protocol Set) | 48 |
| Template 14 | Non-inferiority assessment of anti-Me and anti-Ru antibody seroconversion rates in Coad and Control groups, Differences, Month 4 (Per-Protocol Set) | 49 |
| Template 15 | Non-inferiority assessment of anti-YF antibody seropositivity rate in Coad and Control groups, Difference, Month 4 (Per-Protocol Set) | 49 |
| Template 16 | Anti-CS seropositivity rates and GMTs in Coad and RTS,S groups. Month 4 (Per-Protocol Set) | 49 |

200596 (MALARIA-073) Statistical Analysis Plan Final

| Template 17 | Anti-HBs seropositivity and seroprotection rates and GMTs in Coad and RTS,S groups, Month 4 (Per-Protocol Set) |
|---|---|
| Template 18 | Anti-HBs response to RTS,S/AS01E in Coad and RTS,S groups, GMT ratio, Month 4 (Per-Protocol Set) |
| Template 19 | Anti-Measles seropositivity rates and GMTs in Coad and Control groups, Month 4 (Per-Protocol Set)50 |
| Template 20 | Anti-Rubella seropositivity and seroprotection rates and GMTs in Coad and Control groups, Month 4 (Per-Protocol Set)51 |
| Template 21 | Anti-YF seropositivity rates and GMTs in Coad and Control groups, Month 4 (Per-Protocol Set) |
| Template 22 | Anti-catalase seropositivity rates and GMCs in Coad and Control groups, Month 4 (Per-Protocol Set) |
| Template 23 | Reverse Cumulative Distributions of Anti-CS Titres at Month 4, Coad and RTS,S groups (Per-Protocol Set) |
| Template 24 | Reverse Cumulative Distributions of Anti-Me titres at Month 4,<br>Coad and Control groups (Per-Protocol Set)53 |
| Template 25 | Compliance to data capture per study group (Exposed Set)54 |
| Template 26 | Incidence and nature of solicited and unsolicited symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) |
| Template 27 | Incidence and nature of local solicited and unsolicited symptoms reported for each vaccine over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) |
| Template 28 | Incidence and nature of grade 3 solicited and unsolicited symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) |
| Template 29 | Incidence and nature of local grade 3 solicited and unsolicited symptoms reported for each vaccine over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) |
| Template 30 | Incidence and nature of solicited and unsolicited symptoms considered as causally related over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) |
| Template 31 | Incidence and nature of solicited and unsolicited symptoms with considered causal relationship to vaccination, reported for each vaccine, over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) |

200596 (MALARIA-073) Statistical Analysis Plan Final

| Template 32 | Incidence of solicited local symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) | 61 |
|---|---|---|
| Template 33 | Incidence of solicited local symptoms over 7 days post vaccination (Days 1-7) by dose and overall, by vaccine, per study group (Exposed Set) | 63 |
| Template 34 | Incidence of solicited general symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set) | 66 |
| Template 35 | Maximum temperature reported during the 7-day (Days 1-7) post-vaccination period (overall doses), per study group (Exposed Set) | 69 |
| Template 36 | Maximum temperature reported during the <7>-day (Days 1-<7>) post-vaccination period ( <dose 1="">), per study group (Exposed Set)</dose> | 69 |
| Template 37 | Percentage of subjects reporting unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term over 30 days (Days 1-30) post vaccination, per study group (Exposed Set) | 70 |
| Template 38 | Percentage of subjects reporting Serious Adverse Events (SAEs) classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post vaccination, per study group, Month 4.5 (Exposed Set) | 70 |
| Template 39 | Percentage of subjects with fatal SAEs classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post vaccination, per study group, Month 4.5 (Exposed Set) | 71 |
| Template 40 | Percentage of subjects reporting SAEs with causal relationship to vaccination classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post vaccination, per study group, Month 4.5 (Exposed Set) | 71 |
| Template 41 | Listing of SAEs reported until Month 4.5 visit, per study group (Exposed Set) | 71 |
| Template 42 | Incidence of seizures by diagnostic certainty level within 7 days (1-7) post vaccination overall doses (Diagnostic certainty 1-5), per study group (Exposed Set) | 72 |
| Template 43 | Incidence of seizures by diagnostic certainty level and history of fever within 7 days (1-7) post vaccination overall doses (Diagnostic certainty 1-5), per study group (Exposed Set) | 72 |
| Template 44 | Incidence of seizures by diagnostic certainty level and fever within 7 days (1-7) post vaccination overall doses (Diagnostic certainty 1-5), per study group (Exposed Set) | 73 |

| | 200596 (MALARIA-0<br>Statistical Analysis Plan F | |
|---|---|---|
| Template 45 | Incidence of concomitant medication administered during the <30-day (Days 1-30)> post-vaccination period by dose and overall, per study group (Exposed Set) | .74 |
| Template 46 | Number (%) of subjects with serious adverse events including number of events reported during the study period (Exposed Set) | .74 |
| Template 47 | Solicited and unsolicited symptoms, classified by MedDRA Primary System Organ Class and Preferred Term within the 42- day (Days 1-42) post-vaccination period including number of events - SAE excluded (Exposed Set) | .75 |
| Template 48 | Listing of dropouts due to AEs, SAEs and solicited symptoms (Exposed Set) | .75 |

200596 (MALARIA-073) Statistical Analysis Plan Final

#### LIST OF ABBREVIATIONS

AE Adverse event

ANOVA Analysis of Variance

Anti-CS Antibody to the *Plasmodium falciparum* circumsporozoite (CS) repeat

domain

Anti-HBs Antibody to the hepatitis B surface antigen

Anti-Me Anti-measles antibody

Anti-Ru Anti-rubella antibody

Anti-YF Anti-yellow fever antibody

AS01<sub>E</sub> GSK's proprietary Adjuvant System containing MPL, QS-21

Stimulon<sup>®</sup> and liposome (25 μg MPL and 25 μg QS-21 Stimulon<sup>®</sup>)

CI Confidence interval

Coad Co-administration

CS Circumsporozoite protein of *Plasmodium falciparum* 

eCRF Electronic case report form

ED50 End point Dilution 50

EPI Expanded Program on Immunization

ES Exposed Set

EU/ml ELISA unit per milliliter

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titre

GSK GlaxoSmithKline

ICH International Conference on Harmonization

IDMC Independent Data Monitoring Committee

IU/ml International units per milliliter

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PD Protocol Deviation

200596 (MALARIA-073) Statistical Analysis Plan Final

pIMD Potential immune-mediated disease

PPS Per Protocol Set

RCD Reverse cumulative distribution

RTS,S Particulate antigen, containing both RTS and S (hepatitis B surface

antigen) proteins

RTS,S/AS01<sub>E</sub> GSK Biologicals' candidate *Plasmodium falciparum* malaria vaccine

adjuvanted with GSK Biologicals' proprietary Adjuvant System

AS01<sub>E</sub>

SAE Serious adverse event

SAP Statistical Analysis Plan

SD Standard Deviation

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

YF Yellow fever

200596 (MALARIA-073) Statistical Analysis Plan Final

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|---------------------|
| 09-APR-2018 | Final version | Amendment 1 Final – |
| | | 09-AUG-2016 |

# 2. STUDY DESIGN

Figure 1 Study design



09-APR-2018 

- Experimental design: Phase IIIB, open, randomized, controlled, multi-centric study with three parallel groups.
- Duration of the study: Approximately 33 months per participant in the Coad or the RTS,S group and 36 months in the Control group.
  - Epoch 001: Primary starting at Visit 1 (Screening) and ending at Visit 15 (Month 36).
- Study groups: 3 study groups are defined for the study (Coad group, RTS,S group and Control group). A description of the vaccination, blood sample and visit schedule is provided for each of the study groups in Figure 1.

Table 1 Study groups and epochs foreseen in the study

| Study groups | Number of subjects | Age (Min) | Epoch 001 |
|---------------|--------------------|-----------|-----------|
| Coad group | 233 | 6 months* | X |
| RTS,S group | 233 | 6 months* | Х |
| Control group | 233 | 6 months* | х |

<sup>\*</sup> For clarity this corresponds from the day the child becomes 6 months of age until the day before the child achieves 7 months of age.

Table 2 Study groups and treatment foreseen in the study

| Treatment name | Vaccine/Product name | Study groups | | |
|---|---|---|---|---|
| Treatment name | vaccine/Product name | Coad group | RTS,S group | Control group |
| RTS,S/AS01 <sub>E</sub> | RTS,S | Х | Х | X |
| | AS01E | Х | Х | X |
| Yellow fever | WHO prequalified Yellow<br>Fever | Х | х | Х |
| Measles and<br>Rubella | MR-VAC | Х | х | Х |
| Vitamin A | Vitamin A | Х | Х | X |

MR-VAC: Live attenuated measles virus and rubella virus vaccine (Serum Institute of India)

- Treatment allocation: randomized in a 1:1:1 ratio to each study group.
- Blinding: open

Table 3 Blinding of study epoch

| Study Epoch | Blinding |
|-------------|----------|
| Epoch 001 | open |

- Type of study: self-contained.
- Data collection: Electronic Case Report Form (eCRF).
- Safety monitoring: description of safety monitoring is available in Table 5
- Immunogenicity monitoring:

200596 (MALARIA-073) Statistical Analysis Plan Final

# Table 4 Immunological read-outs

| Blood samp | ling timepoint | | No | | Componento |
|---|---|---|---|---|---|
| Type of contact<br>and timepoint | Sampling<br>timepoint | study group | No.<br>subjects | Component | Components<br>priority rank |
| Visit 2 | Day 0 | Coad group and RTS,S group | 466 | anti-CS | 1 |
| | | Coad group and RTS,S group | 466 | anti-HBs | 2 |
| | | Coad group and Control group | 466 | anti-catalase | 3 |
| Visit 4 | Month 3 | Coad group and Control group | 466 | anti-Me | 1 |
| | | Coad group and Control group | 466 | anti-Ru | 2 |
| Visit 5 | Month 4 | Coad group and RTS,S group | 466 | anti-CS | 1 |
| | | Coad group and RTS,S group | 466 | anti-HBs | 5 |
| | | Coad group and Control group | 466 | anti-catalase | 6 |
| | | Coad group and Control group | 466 | anti-Me | 2 |
| | | Coad group and Control group | 466 | anti-Ru | 3 |
| | | Coad group and Control group | 466 | anti-YF | 4 |

Table 5 Reporting periods for adverse events and serious adverse events

| Visit | 1 | | | 2 | | П | | 3 | | П | | 4 | | | 5 | 6 | 7 | Т | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Children age<br>(Months) | | | | 6 | | | | 7.5 | | | | 9 | | 1 | 10 | 10.5 | 11. | 5 | 12.5 | 13.5 | 27 | 28 | 30 | 31 | 39 | 42 |
| Study Month | | 1 | | M0 | | | | M1.5 | | П | | M3 | | N | VI4 | M4.5 | M5. | 5 | M6.5 | M7.5 | M21 | M22 | M24 | M25 | M33 | M36 |
| | D-28<br>to -1 | | D0 | D6 | D29 | | M1.5 | M1.5<br>+6d | M1.5<br>+29d | | М3 | M3<br>+13d | M3<br>+41d | | | | | | | | | | | | | |
| Solicited local<br>and general AEs | | | Ха | Хa | | | Ха | Ха | | | <b>X</b> a | | | | | | | | | | | | | | | |
| Unsolicited AEs | | | Χb | Χþ | Χþ | | Χp | Χp | Xp | | Χp | Χp | Χp | ) | Χþ | Xb,c | Хс | | Хс | Хс | Χq | Χq | Xe | Xe | | |
| SAEs related to<br>study<br>participation or<br>concurrent GSK<br>medication/vacci<br>ne | | | | | | | | | | | | | | | | | | | | | | | | | | |
| SAEs (All, fatal,<br>related to the<br>investigational<br>vaccine) | | | | | | | | | | | | | | | | | | | | | | | | | | |
| AEs of specific interest** | | | | | | | | | | | | | | | | | | | | | | | | | | |

M: study month; d: day

09-APR-2018 

<sup>\*\*</sup> AEs of specific interest include seizure (occurring within 30 days post-vaccination for vaccine doses administered at 6 and 7.5 months of age [Visits 2 and 3] or 42 days post-vaccination for vaccine doses administered at 9 months of age [Visit 4]), meningitis and pIMDs.

a In the Control group, only solicited general AE will be collected. In the Coad and the RTS,S groups, solicited local and general AEs will be collected.

b Unsolicited AEs will be collected from Visit 2 until 42 days after Visit 4 for children in Coad, RTS,S and Control groups.

c Unsolicited AEs will be collected from Visit 6 until 30 days after Visit 8 only for children from the Control group.

d Unsolicited AEs will be collected over a 30-day follow-up period after vaccination only for children from the Coad and the RTS,S groups.

e Unsolicited AEs will be collected over a 30-day follow-up period after vaccination only for children from the Control group.

## 3. OBJECTIVES

# 3.1. Primary objective

- To demonstrate the non-inferiority of the antibody response to the CS antigen when RTS,S/AS01<sub>E</sub> is co-administered with YF vaccine and a combined measles and rubella vaccine versus RTS,S/AS01<sub>E</sub> administered alone.
  - Criteria for non-inferiority: one month post Dose 3 of RTS,S/AS01<sub>E</sub>, the upper limit (UL) of the 2-sided 95% confidence interval (CI) on the geometric mean titre (GMT) ratio (RTS,S group/Coad group) of the anti-CS, is below a limit of 2.

Refer to Section 4.1 for the definition of the primary endpoints.

## 3.2. Secondary objectives

#### **Immunogenicity**

- To describe the antibody response to the CS antigen when RTS,S/AS01<sub>E</sub> is administered at 6, 7.5 and 9 months of age in co-administration with YF vaccine and a combined measles and rubella vaccine versus RTS,S/AS01<sub>E</sub> administered alone.
- To describe the antibody response to the hepatitis B surface (HBs) antigen when RTS,S/AS01<sub>E</sub> is administered at 6, 7.5 and 9 months of age in co-administration with YF vaccine and a combined measles and rubella vaccine versus RTS,S/AS01<sub>E</sub> administered alone.
- To demonstrate the non-inferiority of the antibody response to the measles vaccine antigen when YF vaccine and a combined measles and rubella vaccine are coadministered with RTS,S/AS01<sub>E</sub> versus administration without RTS,S/AS01<sub>E</sub>.
  - Criteria for non-inferiority: one month post-vaccination with the combined measles and rubella vaccine, the UL of the 95% CI on the difference in seroconversion rates of the anti-measles antibody (anti-Me), is below 10% (Control group minus Coad group).
- To describe the antibody response to the measles vaccine antigen when YF vaccine and a combined measles and rubella vaccine are co-administered with RTS,S/AS01<sub>E</sub> versus administration without RTS,S/AS01<sub>E</sub>.
- To demonstrate the non-inferiority of the antibody response to the rubella vaccine antigen when YF vaccine and a combined measles and rubella vaccine are coadministered with RTS,S/AS01<sub>E</sub> versus administration without RTS,S/AS01<sub>E</sub>.
  - Criteria for non-inferiority: one month post-vaccination with the combined measles and rubella vaccine, the UL of the 95% CI on the difference in seroconversion rates of the anti-rubella antibody (anti-Ru), is below 10% (Control group minus Coad group).

200596 (MALARIA-073) Statistical Analysis Plan Final

- To describe the antibody response to the rubella vaccine antigen when YF vaccine and a combined measles and rubella vaccine are co-administered with RTS,S/AS01<sub>E</sub> versus administration without RTS,S/AS01<sub>E</sub>.
- To demonstrate the non-inferiority of the antibody response to the YF vaccine antigen when YF vaccine and a combined measles and rubella vaccine are coadministered with RTS,S/AS01E versus administration without RTS,S/AS01E.
  - Criteria for non-inferiority: one month post-vaccination with the YF vaccine, the UL of the 95% CI on the difference in seropositivity rates of the anti-yellow fever antibody (anti-YF), is below 10% (Control group minus Coad group).
- To describe the antibody response to the YF vaccine antigen when YF vaccine and a combined measles and rubella vaccine are co-administered with RTS,S/AS01<sub>E</sub> versus administration without RTS,S/AS01<sub>E</sub>.

#### Safety

Evaluation of the safety profile of RTS,S/AS01<sub>E</sub> when administered at 6, 7.5 and 9 months of age in co-administration with YF vaccine and a combined measles and rubella vaccine versus RTS,S/AS01<sub>E</sub> administered alone.

Refer to Section 4.2 for the definition of the secondary endpoints.

# 3.3. Tertiary objective

#### **Immunogenicity**

 To describe the antibody response to the human catalase after administration of a 3dose course of RTS,S/AS01<sub>E</sub>.

Refer to Section 4.3 for the definition of the tertiary endpoint.

#### 4. ENDPOINTS

# 4.1. Primary endpoints

- Non-inferiority of the antibody response to the CS antigen (RTS,S group/Coad group):
  - Anti-CS antibody titres at one month post Dose 3 of RTS, S/AS01<sub>E</sub> (Month 4).

# 4.2. Secondary endpoints

#### **Immunogenicity**

- Antibody response to the candidate vaccine RTS,S/AS01<sub>E</sub> (RTS,S group and Coad group):
  - Anti-CS antibody titres and seropositivity (≥ 1.9 EU/ml) at Day 0 and at one month post Dose 3 of RTS,S/AS01<sub>E</sub> (Month 4).
  - Anti-HBs antibody titres and seroprotection (≥ 10 mIU/ml) at Day 0 and at one month post Dose 3 of RTS,S/AS01<sub>E</sub> (Month 4).
- Non-inferiority of the antibody response to the measles vaccine antigen in the combined measles and rubella vaccine (Control group minus Coad group):
  - Seroconversion for anti-Me at one month post-vaccination with the combined measles and rubella vaccine (Month 4). Seroconversion is defined as children with an anti-Me pre-vaccination titre below 150 mIU/ml and a post-vaccination titre ≥ 150 mIU/ml.
- Antibody response to the measles vaccine antigen in the combined measles and rubella vaccine (Control group and Coad group):
  - Anti-Me antibody titres and seropositivity (≥ 150 mIU/ml) pre-vaccination (Month 3) and one month post-vaccination with the combined measles and rubella vaccine (Month 4).
- Non-inferiority of the antibody response to the rubella vaccine antigen in the combined measles and rubella vaccine (Control group minus Coad group):
  - Seroconversion for anti-Ru at one month post-vaccination with the combined measles and rubella vaccine (Month 4). Seroconversion is defined as children with an anti-Ru pre-vaccination titre below 4 IU/ml and a post-vaccination titre ≥ 4 IU/ml.
- Antibody response to the rubella vaccine antigen in the combined measles and rubella vaccine (Control group and Coad group):
  - Anti-Ru antibody titres and seropositivity (≥ 4 IU/ml) pre-vaccination (Month 3) and one month post-vaccination with the combined measles and rubella vaccine (Month 4).
- Non-inferiority of the antibody response to the YF vaccine antigen (Control group minus Coad group):
  - Seropositivity (≥10 ED50) for anti-YF at one month post-vaccination with the YF vaccine (Month 4).
- Antibody response to the YF vaccine antigen (Control group and Coad group):
  - Anti-YF antibody titres and seropositivity (≥ 10 ED50) one month postvaccination with the YF vaccine (Month 4).

#### Safety

- Solicited local and general AEs.
  - For the Coad and the RTS,S groups, the occurrence of solicited local and general AEs over a 7-day follow-up period (day of administration and 6 subsequent days) after administration of Vitamin A and study vaccines at 6 months of age (Visit 2).
  - For the Control group, the occurrence of solicited general AEs over a 7-day follow-up period (day of administration and 6 subsequent days) after administration of Vitamin A at 6 months of age (Visit 2).
  - For the Coad and the RTS,S groups, the occurrence of solicited local and general AEs over a 7-day follow-up period (day of vaccination and 6 subsequent days) after dose of study vaccines administered at 7.5 months of age (Visit 3).
  - For the Control group, the occurrence of solicited general AEs over a 7-day follow-up period (day of visit and 6 subsequent days) after Visit 3 (7.5 months of age).
  - For all groups, the occurrence of solicited general and local AEs over a 14-day follow-up period (day of vaccination and 13 subsequent days) after dose of study vaccines administered at 9 months of age (Visit 4).

#### Unsolicited AEs.

- For all groups, the occurrence of unsolicited AEs over a 30-day follow-up period (day of administration and 29 subsequent days) after administration of Vitamin A and study vaccines at 6 months of age (Visit 2).
- For the Coad and the RTS,S groups, the occurrence of unsolicited AEs over a 30-day follow-up period (day of vaccination and 29 subsequent days) after dose of study vaccines administered at 7.5 months of age (Visit 3).
- For the Control group, the occurrence of unsolicited AEs over a 30-day follow-up period (day of visit and 29 subsequent days) after Visit 3 (7.5 months of age).
- For all groups, the occurrence of unsolicited AEs over a 42-day follow-up period (day of vaccination and 41 subsequent days) after dose of study vaccines administered at 9 months of age (Visit 4).
- For the Coad and the RTS,S groups, the occurrence of unsolicited AEs over a 30-day follow-up period (day of vaccination and 29 subsequent days) after the booster dose of study vaccine administered at 27 months of age (Visit 10).
- For the Control group, the occurrence of unsolicited AEs over a 30-day follow-up period (day of vaccination and 29 subsequent days) after dose of study vaccines administered at 10.5, 11.5, 12.5 and 30 months of age (Visit 6, 7, 8 and 12).

- SAEs: all, fatal and related SAEs.
  - The occurrence of SAEs occurring within 30 days (day of vaccination and 29 subsequent days) after each administration.
  - The occurrence of SAEs from Screening visit (Visit 1) until Month 4.5.
  - The occurrence of SAEs from Screening visit (Visit 1) until study end (Month 33 for Coad and RTS,S groups and Month 36 for the Control group).
  - The occurrence of pIMDs from Day 0 until Month 4.5.
  - The occurrence of pIMDs from Day 0 until study end (Month 33 for Coad and RTS,S groups and Month 36 for the Control group).
  - The occurrence of meningitis from Day 0 until Month 4.5.
  - The occurrence of meningitis from Day 0 until study end (Month 33 for Coad and RTS,S groups and Month 36 for the Control group).
  - The occurrence of seizure (occurring within 30 days post-vaccination for vaccine doses administered at 6 and 7.5 months of age [Visits 2 and 3] or 42 days post-vaccination for vaccine doses administered at 9 months of age [Visit 4]) from Day 0 until Month 4.5.
  - The occurrence of seizure occurring within 30 days post-vaccination for vaccine doses administered at 6, 7.5 and 27 months of age (Visits 2, 3 and 10 for Coad and RTS,S group) and at 10.5, 11.5, 12.5 and 30 months of age (Visits 6, 7, 8 and 12 for Control group) or 42 days post-vaccination for vaccine doses administered at 9 months of age (Visit 4 for all groups).
  - The occurrence of generalized convulsive seizure occurring within 7 days after vaccines administered at Visit 2 and 3 (Coad and RTS,S groups) and 14 days after vaccines administered at Visit 4 (all groups).

# 4.3. Tertiary endpoints

#### **Immunogenicity**

- Antibody response to component of the candidate vaccine RTS,S/AS01<sub>E</sub> (Coad group and Control group):
  - Anti-catalase antibody concentrations and seropositivity at Day 0 and before administration of RTS,S/AS01<sub>E</sub> (Month 4) for the Control group and at Day 0 and at one month post Dose 3 of RTS,S/AS01<sub>E</sub> (Month 4) for the Coad group.

## 5. ANALYSIS SETS

## 5.1. Definition

#### 5.1.1. Enrolled Set

The enrolled set will include all subjects who signed informed consent.

# 5.1.2. Exposed Set (ES)

The exposed set (ES) will include all subjects who received at least one dose of the study treatment (i.e. receiving at least one dose of study vaccine or Vitamin A). The ES analysis will be performed per treatment actually administered.

# Per-Protocol Set for analysis of immunogenicity (PPS for immunogenicity)

The PPS for analysis of immunogenicity will include all evaluable subjects meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study. Subjects with incomplete vaccination course or blood sampling performed outside the protocol defined windows will be eliminated.

Note that in order to align to ICH terminology the Total Vaccinated Cohort and the According To Protocol cohort have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively.

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set. Time intervals were defined in advance and are stored in the elimination form document (MALARIA-073 (200596) Criteria for Eliminating Subjects from the Analysis (main analysis visit 6) (12-Feb-2017) version 2.5) in eTMF.

# 5.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

# 5.2.2. Elimination from Per-protocol analysis Set (PPS)

# 5.2.2.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions. These apply to the period from Day 0 to Visit 6.

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data |
| 1030 | Study vaccine not administered at all |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol |
| 1050 | Randomization failure |
| 1070 | Vaccination not according to protocol: |
| | Incomplete vaccination course before treatment withdrawal. |
| | Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number). |
| | Administered study vaccine reported as being the correct one but is not compatible with the vaccine regimen associated to the treatment number. |
| 1080 | Vaccine temperature deviation (non GMP use) |
| 1090 | Expired vaccine administered |
| 2010 | Protocol violation (inclusion/exclusion criteria) |
| 2040 | Administration of any medication forbidden by the protocol |
| 2050 | Underlying medical condition forbidden by the protocol |
| 2080 | Subjects did not comply with vaccination schedule |
| 2090 | Subjects did not comply with blood sample schedule |
| 2100 | Serological results not available post-vaccination |
| 2120 | Obvious incoherence or abnormality or error in data |

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

Important protocol deviations not leading to elimination from PPS are defined in MALARIA-073 Protocol Deviation Management Plan.

## 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in Section 11 and will not be repeated below.

All statistical analyses will be performed using SAS 9.2 or later versions.

## 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age, gender, length for age Z-score, and weight for age Z-score) of each cohort (ES and PPS for immunogenicity) will be tabulated per study group.

The mean age at first vaccination [Vitamin A administration for Control group] (in months, 1 decimal digit) (plus range and standard deviation) of the vaccinated subjects, as a whole, and per group, will be calculated.

#### 6.1.2. Additional considerations

Demographic characteristics, cohort description, withdrawal status will be summarized by group using descriptive statistics:

- Frequency tables will be generated for categorical variables such as gender.
- Mean, median, standard deviation, minimum and maximum will be provided for continuous data such as age.
- The withdrawal status will be summarized by group using descriptive statistics.
- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses will be tabulated.
- The numbers of withdrawn subjects will be tabulated according to the main reason for withdrawal.

## 6.2. Exposure

## 6.2.1. Analysis of exposure planned in the protocol

The number and percentage of subjects who received study vaccine doses will be tabulated for each study group (ES).

#### 6.2.2. Additional considerations

Not Applicable.

# 6.3. Efficacy/Effectiveness

#### 6.3.1. Analysis of efficacy planned in the protocol

Not Applicable.

#### 6.3.2. Additional considerations

Not Applicable.

## 6.4. Immunogenicity

# 6.4.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PPS for immunogenicity.

For the primary endpoint, the 95% CIs of the anti-CS GMT ratio between the groups (RTS,S group over Coad group) at one month post Dose 3 of RTS,S/AS01<sub>E</sub> will be calculated. Non-inferiority of anti-CS immune response will be concluded if the UL of this CI is below 2.

For the secondary endpoints, the 95% CIs of the difference in anti-Me, anti-Ru and anti-YF seroconversion/seropositivity rates between the groups (Control group minus Coad group) at one month post-vaccination will be calculated (standardized asymptotic). The seroconversion rate is defined as the percentage of initially seronegative that are seropositive post-vaccination. Non-inferiority will be concluded if the UL of this CI is below 10%.

The percentage of subjects with seropositive levels of anti-CS (proportion of subjects with anti-CS antibody titres  $\geq$  **1.9** EU/ml) with 95% CI will be determined at Day 0 and one month post Dose 3 of RTS,S/AS01<sub>E</sub> in the RTS,S group and Coad group. Antibody titres will be summarized by GMT with 95% CI. Antibody titres at one month post Dose 3 of RTS,S/AS01<sub>E</sub> will also be investigated using reverse cumulative curves.

200596 (MALARIA-073) Statistical Analysis Plan Final

Seroprotection level for anti-HBs with 95% CI will be determined at Day 0 and one month post Dose 3 of RTS,S/AS01<sub>E</sub> in the RTS,S group and Coad group. Anti-HBs titres will be summarized by GMT with 95% CI. Anti-HBs titres one month post Dose 3 of RTS,S/AS01<sub>E</sub> will also be investigated using reverse cumulative curves.

Seropositivity levels of anti-Ru ( $\geq$  4 IU/ml) and seropositivity levels of anti-Me ( $\geq$  150 mIU/ml) with 95% CI will be determined pre-vaccination and one month post-vaccination with the YF vaccine and the combined measles and rubella vaccine in the Control group and Coad group. Antibody titres will be summarized by GMT with 95% CI. Anti-Ru and anti-Me titres at one month post-vaccination with the YF vaccine and the combined measles and rubella vaccine will also be investigated using reverse cumulative curves.

Seropositivity levels of anti-YF ( $\geq$  10 ED50) with 95% CI will be determined one month post-vaccination with the YF vaccine and the combined measles and rubella vaccine in the Control group and Coad group. Antibody titres will be summarized by GMT with 95% CI. Anti-YF titres at one month post-vaccination with the YF vaccine and the combined measles and rubella vaccine will also be investigated using reverse cumulative curves.

For the tertiary endpoints, the anti-catalase concentrations will be summarized by seropositivity and geometric mean concentration with 95% CI at Day 0 (Control and Coad groups), at one month post Dose 3 of RTS,S/AS01<sub>E</sub> in the Coad group and before administration of the first dose of RTS,S/AS01<sub>E</sub> in the Control group.

#### 6.4.2. Additional considerations

Standard data derivation procedures for immunogenicity are available in Section 11 (see Section 11.2.4).

The primary analysis will be based on the PPS cohort for analysis of immunogenicity. If, the percentage of vaccinated subjects with serological results excluded from the PPS cohort for analysis of immunogenicity is 5% or more, a second analysis based on the ES will be performed to complement the PPS analysis.

Statistical methods for Geometric Mean Titres/Concentrations and GMT ratio

#### Within group assessment

GMTs and GMCs and associated two-sided 95% CIs will be computed for each group and for each strain at each available immunogenicity monitoring (see Section 6.4–Immunogenicity monitoring). The 95% CI for the mean of log-transformed titre (or concentration) will be first obtained assuming that log-transformed titres (or concentrations) are normally distributed with unknown variance. Logarithmic transformations use base 10. The 95% CI for the GMT (or GMC) will then be obtained by exponential transformation (base 10) of the 95% CI for the mean of the log-transformed titres (or concentrations).

200596 (MALARIA-073) Statistical Analysis Plan Final

#### Between group assessment

The group GMT ratio (RTS,S group over Coad group) of anti-CS at one month post Dose 3 of RTS,S/AS01<sub>E</sub> will be obtained using an ANOVA model on the logarithm-transformed titres. The ANOVA model will include the study group as fixed effect. The GMT ratio and its two-sided 95% CI will be derived as exponential-transformation (base 10) of the corresponding group contrast in the model.

#### Reverse cumulative distribution curves

Reverse cumulative distribution (RCD) curves for antibody titres will be plotted: the x-axis represents the antibody titres value (log-10 scale), while the y-axis the percentage of subjects having a log-transformed antibody value greater or equal to the corresponding x-value. RCD curves analysis is performed by study group for the following immunogenicity monitoring:

- one month post Dose 3 of RTS,S/AS01E for anti-CS and anti-HBs titres
- one month post-vaccination with the YF vaccine and the combined measles and rubella vaccine for anti-Me, anti-Ru and anti-YF titres

<u>Statistical methods for seropositivity/seroprotection rates and for seroconversion/seropositivity rates differences</u>

The percentage of subjects seropositive/seroprotected and associated two-sided 95% Clopper-Pearson confidence intervals (CIs) will be computed by vaccine group for each strain at each available immunogenicity monitoring. In addition, differences in percentages (for seroconversion rates of anti-Me and anti-Ru and for the seropositivity rate of anti-YF at one month post-vaccination) between the groups (Control group minus Coad group) will be calculated and the associated confidence interval for the difference will be constructed using the method of Miettinen and Nurminen.

## 6.5. Analysis of safety

## 6.5.1. Analysis of safety planned in the protocol

The primary analysis will be based on the ES.

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the solicited follow-up period [7 days post Dose 1, post Dose 2 and 14 days post Dose 3]will be tabulated with exact 95% CI after each vaccine dose and overall. The percentage of doses followed by at least one local AE (solicited and unsolicited), by at least one general AE (solicited and unsolicited) and by any AE will be tabulated for the overall vaccination course, with exact 95% CI. Similar tables will be generated for Grade 3 AEs and AEs considered as causally related to vaccination.

The percentage of subjects reporting each individual solicited local and general AE during the solicited follow-up period will be tabulated with exact 95% CI. The percentage of doses followed by each individual solicited local and general AE will be tabulated for each dose and for the overall vaccination course, with exact 95% CI. Similar tables will be generated for Grade 3 AEs, causal events and for fever, temperature in 0.5°C increments.

The proportion of subjects reporting an AE (unsolicited) until 30 days (Days 0-29) post each dose of RTS,S/AS01<sub>E</sub>, classified by the Medical Dictionary for Regulatory Activities (MedDRA) preferred term level will be tabulated with exact 95% CI. The proportion of subjects reporting an AE (unsolicited) until 42 days (Days 0-41) after the administration of the YF vaccine and the combined measles and rubella vaccine (restricted to the Coad group and Control group), classified by the MedDRA preferred term level will be tabulated with exact 95% CI. Similar tables will be generated for Grade 3 AEs and AEs considered as causally related to vaccination.

The proportion of subjects reporting an SAE (all, fatal, related) occurring within 30 days (day of vaccination and 29 subsequent days) after each visit where a study product is potentially administered, classified by the MedDRA preferred term level will be tabulated with exact 95% CI.

200596 (MALARIA-073) Statistical Analysis Plan Final

The proportion of subjects reporting an SAE (all, fatal, related) from Day 0 to Month 4.5 and over the whole study duration (Day 0 to Month 33 for Coad and RTS,S groups and Month 36 for the Control group), classified by the MedDRA preferred term level will be tabulated with exact 95% CI.

The proportion of subjects reporting an AEs of specific interest (pIMDs, meningitis and seizures) from Day 0 to Month 4.5 and over the whole study duration (Day 0 to Month 33 for Coad and RTS,S groups and Month 36 for the Control group), classified by the MedDRA preferred term level will be tabulated with exact 95% CI.

For generalized convulsive seizures occurring within 7 days after vaccines administered at Visit 2 and 3 (Coad and RTS,S groups) and 14 days after vaccines administered at Visit 4 (all groups) an analysis will be performed based on the Brighton Collaborations guidelines [Bonhoeffer, 2004]. This includes descriptive tables of the time relationship of seizures to vaccination, the duration of seizures and the level of diagnostic certainty.

#### 6.5.2. Additional considerations

Standard data derivation procedures for safety are available in Section 11 (see Section 11.2.5).

Note that the study will be converted in cDISC. Accordingly Day 0-Day N will be replaced by Day 1-Day N+1 for the statistical analysis.

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited AEs will be provided. Solicited AEs will be coded by MedDRA as per the following codes:

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain at injection site | 10022086 | Injection site pain |
| Redness at injection site | 10022098 | Redness at injection site |
| Swelling at injection site | 10053425 | Swelling at injection site |
| Drowsiness | 10013649 | Drowsiness |
| Fever | 10016558 | Fever |
| Irritability/Fussiness | 10057224 | Irritability post vaccinal |
| Loss of appetite | 10003028 | Appetite lost |
| Measles-like rash | 10027022 | Measles-like rash |

Cases of measles and rubella will be listed.

#### 6.5.2.1. Concomitant Medication and Concomitant Vaccination

Medications will be coded using the GSKDRUG dictionary.

The frequencies and percentages of subjects reporting antipyretic medications will be tabulated by vaccine group for each study dose and across doses. All concomitant medication will be provided in individual listings.

Antipyretics will be further considered prophylactic when administered in the absence of ANY symptom and in anticipation of a reaction to the vaccination.

Concomitant vaccinations administered in the period starting seven days before the first dose of study vaccine and ending at Visit 5 (Month 4) will be listed.

## 7. ANALYSIS INTERPRETATION

Except for analyses on objectives with a pre-defined success criterion (see Section 3), comparative analyses will be descriptive with the aim to characterize the difference in immunogenicity and safety between groups.

## 8. CONDUCT OF ANALYSES

# 8.1. Sequence of analyses

| Descriptio<br>n | Analysi<br>s ID | Disclosure Purpose (CTRS=publi c posting, SR=study report, internal) | Dry<br>run<br>review<br>neede<br>d<br>(Y/N) | Study Headline Summary (SHS)requirin g expedited communicatio n to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final<br>analysis | E1_01 | SR, CTRS | Y | Yes | TFL_TOC_MAL<br>-073 |
| Primary<br>Epoch<br>Analysis | E1_02 | SR, CTRS | Y | Yes | TFL_TOC_MAL<br>-073 |

The primary analysis will be performed on data collected up to and including 42 days post-measles/rubella/YF vaccination and will include all immunogenicity data (primary secondary and tertiary endpoints) and safety data (secondary endpoints) up to Month 4.5 (Visit 6). A clinical study report will be written after this analysis.

An analysis with remaining safety data will be performed when all data up to and including the Month 33 for Coad and RTS,S groups (Visit 14) and Month 36 for the Control group (Visit 15) will be available. Additional safety information will be added to the clinical study report prepared after Visit 6.

# 8.2. Statistical considerations for interim analyses

No interim analyses are planned.

#### 9. CHANGES FROM PLANNED ANALYSES

The seropositivity threshold for anti-CS has been updated from 0.5 EU/ml to 1.9 EU/ml.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analysis and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The mock tables referred under column named 'layout' can be found in Section 13 of this SAP.

The following group names will be used in the TFLs, to be in line with the T-domains:

| Group<br>order in<br>tables | Group label in tables | Group definition for footnote | Pooled<br>Groups label<br>in tables | Pooled<br>definition<br>for footnote |
|---|---|---|---|---|
| 1 | Coad | Group receiving co-<br>administration<br>regimen of<br>RTS,S/AS01 <sub>E</sub> , YF<br>vaccine and a<br>combined measles and<br>rubella vaccine | NA | NA |
| 2 | RTS,S | Group receiving regimen of RTS,S/AS01 <sub>E</sub> vaccine | NA | NA |
| 3 | Control | Group receiving regimen of YF vaccine and a combined measles and rubella vaccine | NA | NA |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper: Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890]. The standardised asymptotic method used is the method six.

#### 11.1.1. Other references

Bonhoeffer J, Menkes J, Gold MS et al. Generalized convulsive seizure as an adverse event following immunization: case definition and guidelines for data collection, analysis and presentation. *Vaccine*. 2004; 22:557-562.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day & month are missing, 30June is used.
- The onset day for a safety event is the number of days between the last study vaccination and the onset/start date of the event (onset date last study vaccination+1). This is 1 for an event starting on the same day as a vaccination.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore duration is 1 day for an event starting & ending on the same day.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which
  vaccination occurred. More specifically dose 1 refers to all vaccines administered at
  the first vaccination visit while dose 2 corresponds to all vaccinations administered
  at the second vaccination visit even if this is the first time a product is administered
  to the subject.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (eg 3<sup>rd</sup> study dose), the relative dose of the event will be study dose associated to the subsequent study dose (eg dose 3).
  - The number of doses for a product is the number of time the product was administered to a subject.
  - The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

## 11.2.3. Demography

Age: Age at the reference activity, computed as the number of days between the date
of birth and the reference activity and converted in months (= days \*12 /365.25)
(keeping 1 decimal digit).

## 11.2.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or nonevaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.
- The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations (base 10). Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT calculation. The cut-off value is defined by the laboratory before the analysis.
- A subject seropositive for anti-CS antibody will be a subject whose antibody titre
  will be greater than or equal to the cut-off value (anti-CS ≥ 1.9 EU/ml).
- A subject seropositive for anti-HBs antibody will be a subject whose antibody titre will be greater than or equal to the cut-off value (anti-HBs ≥ 6.2 mIU/ml).
- Seroprotection rate for anti-HBs antibody is defined as the percentage of subjects with antibody titres greater than or equal to 10 mIU/ml (anti-HBs ≥ 10 mIU/ml).

- Seroconversion rate for anti-Me is defined as the percentage of children with an anti-Me pre-vaccination titre below 150 mIU/ml and a post-vaccination titre ≥ 150 mIU/ml (i.e. the subject is seropositive post-vaccination and seronegative pre-vaccination for anti-Me).
- Seroconversion rate for anti-Ru is defined as the percentage of children with an anti-Ru pre-vaccination titre below 4 IU/ml and a post-vaccination titre ≥ 4 IU/ml (i.e. the subject is seropositive post-vaccination and seronegative pre-vaccination for anti-Ru).
- Seroprotection rate for anti-Ru antibody is defined as the percentage of subjects with antibody titres greater than or equal to 10 IU/ml (anti-Ru ≥ 10 IU/ml).
- A subject seropositive for anti-YF antibody will be a subject whose antibody titre
  will be greater than or equal to the cut-off value (anti-YF ≥ 10 ED50).
- A subject seropositive for anti-catalase antibody will be a subject whose antibody concentration is greater than or equal to 65 ng/ml.
- The assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'cut\_off', numerical immuno result is derived from a character field (rawres):
  - If rawres is 'NEG' or '-' or '(-)', numeric result= cutt\_off/2,
  - if rawres is 'POS' or '+' or '(+)', numeric result = cut\_off,
  - if rawres is '< value' and value<=cut off, numeric result =cut off/2,</li>
  - if rawres is '< value' and value>cut off, numeric result =value,
  - if rawres is '> value' and value<cut off, numeric result =cut off/2,</li>
  - if rawres is '> value' and value>=cut off, numeric result =value,
  - if rawres is '<= value' or '>= value' and value<cut\_off, numeric result</li>
     ecut\_off/2,
  - if rawres is '<= value' or '>= value' and value>=cut off, numeric result =value,
  - if rawres is a value < cut off, numeric result = cut off/2,</li>
  - if rawres is a value >= cut\_off, numeric result = rawres,
  - if rawres is a value >= cut off, numeric result = rawres,
  - else numeric result is left blank.
  - All CI computed will be two-sided 95% CI.

#### 11.2.5. Safety

- For a given subject and the analysis of solicited symptoms, missing or non-evaluable
  measurements will not be replaced. Therefore the analysis of the solicited symptoms
  based on the Exposed Set will include only vaccinated subjects for doses with
  documented safety data (i.e., symptom screen completed). More specifically the
  following rules will be used:
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
  - Subjects who documented the presence of a solicited symptom and fully or
    partially recorded daily measurement over the solicited period will be included
    in the summaries at that dose and classified according to their maximum
    observed daily recording over the solicited period.
  - Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for other symptoms).
  - Doses without symptom sheets documented will be excluded.
- For analysis of unsolicited adverse events, such as serious adverse events or adverse
  events by primary MedDRA term, and for the analysis of concomitant medications,
  all vaccinated subjects (or receiving Vitamin A) will be considered. Subjects who did
  not report the event or the concomitant medication will be considered as subjects
  without the event or the concomitant medication respectively.
- The maximum intensity of local injection site redness/swelling will be coded as follows:

| Grade | Redness/swelling |
|-------|----------------------|
| 0 | Absent |
| 1 | > 0 mm and < 5<br>mm |
| 2 | ≥ 5 mm and ≤ 20 mm |
| 3 | > 20 mm |
• For the analysis, temperatures will be coded as follows:

| Grade | Temperature |
|-------|---------------------|
| 0 | <37.5°C |
| 1 | ≥ 37.5°C - ≤ 38.0°C |
| 2 | > 38.0°C - ≤ 39.0°C |
| 3 | > 39.0°C |

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per<br>subject for Vaccination phase | N used for deriving % per dose for Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom | All subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited<br>symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

200596 (MALARIA-073) Statistical Analysis Plan Final

# Number of decimals displayed:

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median, SD | 1 |
| Immunogenicity | GMT/C, including LL & UL of CI | 1 |
| Immunogenicity | Ratio of GMT, including LL & UL of CI | 2 |
| All summaries, | % of count, including LL & UL of | 1 |
| Reactogenicity | CI | |
| All summaries | % of difference, including LL & UL of CI | 2 |

# 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Table 6 Safety Sets

| PD code | PD Description | Study<br>Objective/<br>Period | All Exposed Set |
|---|---|---|---|
| | Exclusion code | | EXPFL |
| 1030 | Study vaccine not administered AT ALL | All Study | EXC |
| 900 | Invalid inform<br>consent or fraud<br>data | | EXC |

EXC = excluded from this analysis set.

Table 7 Immunogenicity Sets

| PD code | PD Description | Study<br>Objective/<br>Period | All Exposed | PPS |
|---|---|---|---|---|
| | Exclusion code | | EXPFL | PPSFL |
| 1030 | Study vaccine not<br>administered AT ALL | All Study | EXC | EXC |
| 900 | Invalid inform consent or fraud data | | EXC | EXC |
| 1040 | Administration of forbidden vaccine | | | EXC |
| 1050 | Randomization failure | | | EXC |
| 1070 | Wrong replacement of study vaccine administered | | | EXC |
| 1070 | Administered study vaccine reported as correct but not compatible with regimen associated to treatment number | | | EXC |
| 1070 | Incomplete vaccination course | | | EXC |
| 1080 | Administration of<br>temperature-<br>deviated vaccine | | | EXC |
| 1090 | Administration of expired vaccine | | | EXC |
| 2010 | Subject did not meet entry criteria | | | EXC |
| 2040 | Administration of forbidden medication | | | EXC |
| 2050 | Underlying medical condition forbidden by the protocol | | | EXC |

200596 (MALARIA-073) Statistical Analysis Plan Final

| PD code | PD Description | Study<br>Objective/<br>Period | All Exposed | PPS |
|---|---|---|---|---|
| | Exclusion code | | EXPFL | PPSFL |
| 2080 | Did not comply with<br>study vaccination<br>schedule | | | EXC |
| 2090 | Did not comply with blood draw schedule | | | EXC |
| 2100 | Serological results are not available | | | EXC |
| 2120 | Obvious deviation from Laboratory Manual or error in laboratory data | | | EXC |
| 2120 | Incoherence between CRF and CLS database in terms of sample availability (e.g. sample not collected but result is available) | | | EXC |
| 2120 | Label error of blood<br>samples that could<br>not be resolved | | | EXC |

PPS=Per Protocol Set; EXC = excluded from this analysis set

# 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following drafted study specific mocks will be used.

The data display, title and footnote is for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC. These templates were copied from MALARIA-063 and additional tables required for public disclosure were added.

Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment.

Template 1 Number of subjects enrolled by center, per study group (Exposed Set)

| | | Coad N = | | RTS,S N = | | Control N = | | Total N = | |
|---|---|---|---|---|---|---|---|---|---|
| Center | | n | % | n | % | n | % | n | % |
| PPD | (Ghana) | | | | | | | | |
| PPD | (Ghana) | | | | | | | | |

Coad =

RTS,S =

Control =

N = Number of subjects

n = Number of subjects enrolled by center

Center = GSK Biologicals assigned center number

% = n / Number of subjects with available results x 100

Template 2 Number of enrolled subjects by country (All Enrolled Set)

| | Coad<br>N = | RTS,S<br>N = | Control<br>N = | Total<br>N = |
|---------|-------------|--------------|----------------|--------------|
| Country | N | n | n | n |
| Ghana | | | | |

Coad =

RTS.S =

Control =

N = number of subjects

n= number of enrolled subjects included in each group or in total

Template 3 Number of enrolled subjects by age category (All Enrolled Set)

| | | Coad<br>N = | RTS,S<br>N = | Control<br>N = | Total<br>N = |
|---|---|---|---|---|---|
| Characteristics | Categories | n | n | n | n |
| Age category | Infants and toddlers (28 days- | | | | |
| | 23 months) | | | | |

Coad =

RTS.S =

Control =

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = <describe missing>

200596 (MALARIA-073) Statistical Analysis Plan Final

# Template 4 Consort, per study group (Month 4.5)(all screened set)

| | Total | Coad | RTS,S | Control |
|---|---|---|---|---|
| Screened | | | | |
| Reasons for not being vaccinated | | | | |
| Did not meet eligibility criteria | | | | |
| Migrated/Lost to FU before first vaccination | | | | |
| Other | | | | |
| Protocol violation | | | | |
| Vaccinated (at least one vaccination) | | | | |
| Reasons for incomplete vaccination course | | | | |
| Other | | | | |
| Protocol violation | | | | |
| Serious adverse event | | | | |
| Subjects with full vaccination course | | | | |
| Reasons for elimination from PPS for immunogenicity | | | | |
| Serological results not available | | | | |
| Administration of concomitant vaccination | | | | |
| Wrong replacement | | | | |
| Inclusion criteria not met | | | | |
| Out of interval | | | | |
| PPS for immunogenicity | | | | |

Coad = RTS,S =

Control =

Template 5 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal until Month 4.5, per study group (Exposed Set)

| | Coad | RTS,S | Control | Total |
|---|---|---|---|---|
| Number of subjects vaccinated | | | | |
| Number of subjects completed | | | | |
| Number of subjects withdrawn | | | | |
| Reasons for withdrawal : | | | | |
| Serious Adverse Event | | | | |
| Non-Serious Adverse Event | | | | |
| Protocol violation | | | | |
| Consent withdrawal (not due to an adverse event) | | | | |
| Migrated/moved from study area | | | | |
| Lost to follow-up (subjects with incomplete | | | | |
| vaccination course) | | | | |
| Lost to follow-up (subjects with complete | | | | |
| vaccination course) | | | | |
| Sponsor study termination | | | | |
| Others | | | | |

Coad =

RTS,S =

Control =

Vaccinated = number of subjects who were vaccinated in the study Completed = number of subjects who completed Month 4.5 visit Withdrawn = number of subjects who did not come for the last visit

# Template 6 Deviations from specifications for age and intervals between study visits (Exposed Set)

| | | Age | Dose1-Dose2 | Dose1-Dose3 | Dose1-<br>PI(D30) | Dose2-<br>PII(D90) | Dose3-<br>PIII(D210) | Dose1-<br>PIII(D420) |
|---|---|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Protocol | Protocol | Protocol | Protocol |
| | | from 50 to | from 60 to 70 | | from 30 to 40 | from 30 to 40 | from 30 to 40 | from 420 to |
| | | 70 year | days | 194 days | days | days | days | 440 days |
| 10-<br>PLAIN | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| 30-<br>PLAIN | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| 10-AL | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| 30-AL | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| 10-<br>AS01E | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| 30-<br>AS01E | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| 10-<br>AS04C | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| 30-<br>AS04C | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |
| Placebo | N | | | | | | | |
| | n | | | | | | | |
| | % | | | | | | | |
| | range | | | | | | | |

<sup>10-</sup>PLAIN = 3 doses of non-adjuvanted vaccine containing 10 mcg of each antigen

<sup>30-</sup>PLAIN = 3 doses of non-adjuvanted vaccine containing 30 mcg of each antigen

<sup>10-</sup>AL = 3 doses of aluminium adjuvanted vaccine containing 10 mcg of each antigen

<sup>30-</sup>AL = 3 doses of aluminium adjuvanted vaccine containing 30 mcg of each antigen

<sup>10-</sup>AS01E = 2 doses of AS01e adjuvanted vaccine containing 10 mcg of each antigen and 1 dose of saline solution

<sup>30-</sup>AS01E = 2 doses of AS01e adjuvanted vaccine containing 30 mcg of each antigen and 1 dose of saline solution

200596 (MALARIA-073) Statistical Analysis Plan Final

10-AS04C = 2 doses of AS04c adjuvanted vaccine containing 10 mcg of each antigen and 1 dose of saline solution 30-AS04C = 2 doses of AS04c adjuvanted vaccine containing 30 mcg of each antigen and 1 dose of saline solution Placebo = 3 doses of saline solution

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

PI(D30) = One month post-dose 1 blood sample time point - Day 30 (visit 3)

PII(D90) = One month post-dose 2 blood sample time point - Day 90 (visit 6)

PIII(D210) = One month post-dose 3 blood sample time point - Day 210 (visit 9)

PIII(D420) = Eight months post-dose 3 blood sample time point - Day 420 (visit 10)

Template 7 Number of subjects at each visit and list of withdrawn subjects until Month 4.5, per study group (Exposed Set)

| Group | VISIT | N | Withdrawn Subject numbers | Reason for withdrawal |
|---------|-----------|---|---------------------------|-----------------------|
| Coad | SCREENING | | | |
| | VISIT2 | | | |
| | VISIT3 | | | |
| | VISIT4 | | | |
| | VISIT5 | | | |
| | VISIT6 | | | |
| RTS,S | SCREENING | | | |
| - | VISIT2 | | | |
| | VISIT3 | | | |
| | VISIT4 | | | |
| | VISIT5 | | | |
| | VISIT6 | | | |
| Control | SCREENING | | | |
| | VISIT2 | | | |
| | VISIT3 | | | |
| | VISIT4 | | | |
| | VISIT5 | | | |
| | VISIT6 | | | |

Coad =

RTS,S =

Control =

N = Number of subjects who are still in the study up to the visit

Withdrawn = Subject who did not return after the visit

200596 (MALARIA-073) Statistical Analysis Plan Final

# Template 8 Number and percentage of subjects who received study vaccine doses by vaccine, per study group (Exposed Set)

| | CoadRT | S,SA | Coa | d | Coad Y | ellow | RTS | ,S | RTS | ,S | RTS,S Y | ellow | Contro | ol |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | S01E | N = | Measles | Measles and | | fever N = | | RTS,SAS01E | | Measles and | | fever N = | | S01 |
| | | | Rubella | Rubella N = | | | | N = | | Rubella N = | | | EN= | • |
| Total<br>number of<br>doses<br>received | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| 0 | | | | | | | | | | | | | | |
| 1 | | | | | | | | | | | | | | |
| 2 | | | | | | | | | | | | | | |
| 3 | | | | | | | | | | | | | | |
| Any | | | | | | | | | | | | | | |

| | Cont<br>Measles<br>Rubella | and | Control<br>Yellow fever<br>N = | |
|---|---|---|---|---|
| Total number of doses received | n | % | n | % |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |
| Any | | | | |

Coad =

RTS,S =

Control =

N = number of subjects in each group included in the considered cohort n/% = number/percentage of subjects receiving the specified total number of doses Any = number and percentage of subjects receiving at least one dose

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 9 Number of subjects enrolled into the study as well as the number excluded from PPS analyses with reasons for exclusion, per study group (all enrolled set)

| | | Total | | | Coad | | RTS,S | Control | |
|---|---|---|---|---|---|---|---|---|---|
| Title | n | s | % | n | s | n | s | n | s |
| Total cohort | | | | | | | | | |
| Study vaccine dose not administrated but subject number allocated ( code 1030 ) | | | | | | | | | |
| Exposed Set | | | | | | | | | |
| Administration of vaccine(s) forbidden in the protocol ( code 1040 ) | | | | | | | | | |
| Randomisation failure ( code 1050 ) | | | | | | | | | |
| Protocol violation (inclusion/exclusion criteria) ( code 2010 ) | | | | | | | | | |
| Non compliance with vaccination schedule (including wrong and unknown dates) (code 2080) | | | | | | | | | |
| Essential serological data missing ( code 2100 ) | | | | | | | | | |
| PPS for immunogenicity | | | | | | | | | |

Coad =

RTS,S =

Control =

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

% = percentage of subjects in the considered PPS relative to the ES

200596 (MALARIA-073) Statistical Analysis Plan Final

# Template 10 Summary of demographic characteristics at baseline, per study group (Exposed Set)

| | | Coad N | = | RTS,S N | <b>V</b> = | Control | N = | Total N = | |
|---|---|---|---|---|---|---|---|---|---|
| Characteristics | Parameters | Value or n | % | Value or n | % | Value or n | % | Value or n | % |
| | or | | | | | | | | |
| | Categories | | | | | | | | |
| Age at first | Mean | | | | | | | | |
| vaccination in | SD | | | | | | | | |
| months | Median | | | | | | | | |
| | Minimum | | | | | | | | |
| | Maximum | | | | | | | | |
| Gender | Female | | | | | | | | |
| | Male | | | | | | | | |
| Length for age z- | Mean | | | | | | | | |
| score [HAZ] | SD | | | | | | | | |
| | Minimum | | | | | | | | |
| | Maximum | | | | | | | | |
| | Missing | | | | | | | | |
| Weight for age z- | Mean | | | | | | | | |
| score [WAZ] | SD | | | | | | | | |
| | Minimum | | | | | | | | |
| | Maximum | | | | | | | | |
| | Missing | | | | | | | | |

Coad =

RTS,S =

Control =

N = number of subject number

n = number of subject number in a given category

Value = value of the considered parameter

% = n / Number of subject number with available results x 100

Template 11 Minimum and maximum activity dates, per study group (Exposed Set)

| Group | Activity number | Activity<br>Description | Minimum<br>date | Maximum<br>date |
|---|---|---|---|---|
| each | each | | | |
| group | activity | | | |

Coad =

RTS,S =

Control =

# Template 12 Eligibility (Total cohort) (all screened set)

| Eligibility criteria | N | % |
|---|---|---|
| A male or female infant aged between 8 and 12 weeks inclusive at the time of first | | |
| vaccination | | |
| Any other findings that would increase the risk of having an adverse outcome from | | |
| participation | | |
| Any other findings that would result in data collected being incomplete or of poor quality | | |
| Born after a normal gestation period of 36 to 42 weeks inclusive | | |
| Healthy subjects as established by medical history and clinical examination before study | | |
| entry | | |
| Laboratory screening tests out of range (see protocol) | | |
| Previous vaccination with diphtheria, tetanus, pertussis (whole-cell or acellular), | | |
| Haemophilus influenzae type b, Streptococcus pneumoniae, hepatitis B vaccine or | | |
| rotavirus vaccines. | | |
| Serious acute or chronic illness determined by clinical or physical exam and lab | | |
| screening tests | | |
| Subjects whom parent(s)/LAR(s) can and will comply with the requirements of the | | |
| protocol | | |

N = Number of times each eligibility criterion was reported as a reason for a subject failing screening

Note: Subjects could fail multiple eligibility criteria. Therefore, the sum of N in this table is greater than the number of subjects that were screening failures due to not meeting the eligibility criteria

LAR: Legally Acceptable Representative

ICF: Informed Consent Form

Template 13 Primary objective assessment: Non-inferiority assessment of anti-CS antibody response to RTS,S/AS01E in Coad and RTS,S groups, GMT ratio, Month 4 (Per-Protocol Set)

| | | | | GMT rat | io (RTS, | 3 / Coad) | |
|----------|---|-------|---|---------|----------|-----------|----|
| | F | RTS,S | | Coad | | 95% CI | |
| Antibody | N | GMT | N | GMT | Value | LL | UL |
| Anti-CS | | | | | | | |

RTS,S =

Coad =

GMT = geometric mean antibody titre

N = Number of subjects with post-vaccination results available

95% CI = 95% confidence interval for the GMT ratio (Anova model - pooled variance); LL = lower limit, UL = upper limit PIII(M4) = Post Dose 3, Month 4

# Template 14 Non-inferiority assessment of anti-Me and anti-Ru antibody seroconversion rates in Coad and Control groups, Differences, Month 4 (Per-Protocol Set)

| | | | | Difference in seroconversion ra<br>(Group 1 minus Group 2) | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % CI | | | |
| Antibody | Group 1 | 1 N % Group 2 N % | | | Difference | % | LL | UL |
| Anti-Me | Control | | Coad | | Control - Coad | | | |
| Anti-Ru | Control | | Coad | | Control - Coad | | | |

Control =

Coad =

N = number of subjects with available results

% = percentage of subjects with Anti-Me/Anti-Ru titre >= . MIU-ML post-vaccination and < .MIU-ML pre-vaccination 95% CI = 95% Standardized asymptotic confidence interval; LL = lower limit, UL = upper limit

PIII(M4) = Post Dose 3, Month 4

# Template 15 Non-inferiority assessment of anti-YF antibody seropositivity rate in Coad and Control groups, Difference, Month 4 (Per-Protocol Set)

| | | | | | | | Difference in seropositivity rate<br>(Group 1 minus Group 2) |
|---|---|---|---|---|---|---|---|
| | | | | | | | 95 % C |
| Group 1 | N | % | Group 2 | N | % | Difference | Difference % LL U |
| Control | | | Coad | | | Control - Coad | |

Control =

Coad =

N = number of subjects with available results

% = percentage of subjects with Anti-YF titre >= . MIU-ML

95% CI = 95% Standardized asymptotic confidence interval; LL = lower limit, UL = upper limit

PIII(M4) = Post Dose 3, Month 4

Template 16 Anti-CS seropositivity rates and GMTs in Coad and RTS,S groups, Month 4 (Per-Protocol Set)

| | | | | >= 1.9 EU/ml | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | 6 CI | 95% CI | | | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-CS | RTS,S | Pre | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | |
| | Coad | Pre | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | |

RTS,S =

Coad =

GMT = geometric mean antibody titre calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

MIN/MAX = Minimum/Maximum

Pre = Day 0

PIII(M4) = Post Dose 3, Month 4

# Template 17 Anti-HBs seropositivity and seroprotection rates and GMTs in Coad and RTS,S groups, Month 4 (Per-Protocol Set)

| >= 6.2 | | | | | = 6.2 | mIU/mL >= | | | >= 10 mIU/mL | | | GMT | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% CI | | | 95% CI | | 95% CI | | | | | | |
| Antibody | Group | Timing | N | n | % | LL | UL | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-HBs | Coad | Pre | | | | | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | | | | | |
| | RTS,S | Pre | | | | | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | | | | | |

RTS,S = Coad =

GMT = geometric mean antibody titre calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

MIN/MAX = Minimum/Maximum

Pre = Day 0

PIII(M4) = Post Dose 3, Month 4

# Template 18 Anti-HBs response to RTS,S/AS01E in Coad and RTS,S groups, GMT ratio, Month 4 (Per-Protocol Set)

| | | | | | ( | GMT rat | io | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | 95% | 6 CI |
| Group description | N | Group<br>description | N | GMT | Ratio order | Value | LL | UL |
| RTS,S | | Coad | | | RTS,S /Coad | | | |

RTS,S =

Coad =

GMT = geometric mean antibody titer

N = Number of subjects with post-vaccination results available

95% CI = 95% confidence interval for the GMC ratio (Anova model - pooled variance with more than 2 groups);

LL = lower limit,

UL = upper limit

Template 19 Anti-Measles seropositivity rates and GMTs in Coad and Control groups, Month 4 (Per-Protocol Set)

| | | | | | >= 150 | mIU/m | nl | | GMT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 9: | 5% CI | | 9! | % CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti- | Coad | Pre | | | | | | | | | | |
| Measles | | | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | |
| | Control | Pre | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | |

Control =

Coad =

GMT = geometric mean antibody titre calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

MIN/MAX = Minimum/Maximum

PRE = Month 3

PIII(M4) = Post Dose 3, Month 4

# Template 20 Anti-Rubella seropositivity and seroprotection rates and GMTs in Coad and Control groups, Month 4 (Per-Protocol Set)

| | | | | | >= 4 | IU/m | I | | >= 10 | IU/m | | | GMT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 959 | % CI | | | 95% | 6 CI | | 95 | % CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-Ru | Coad | Pre | | | | | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | | | | | |
| | Control | Pre | | | | | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | | | | | |

Control =

Coad =

GMT = geometric mean antibody titre calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

MIN/MAX = Minimum/Maximum

PRE = Month 3

PIII(M4) = Post Dose 3, Month 4

# Template 21 Anti-YF seropositivity rates and GMTs in Coad and Control groups, Month 4 (Per-Protocol Set)

| | | | | | >= 10 | ED50 | | | GMT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | 6 CI | | 95% | 6 CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-YF | Coad | PIII(M4) | | | | | | | | | | |
| | Control | PIII(M4) | | | | | | | | | | |

Control =

Coad =

GMT = geometric mean antibody titre calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

MIN/MAX = Minimum/Maximum

PIII(M4) = Post Dose 3, Month 4

Template 22 Anti-catalase seropositivity rates and GMCs in Coad and Control groups, Month 4 (Per-Protocol Set)

| | | | | | >= 65 | ng/ml | | | GMC | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI | | 95 | % CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-<br>catalase | Coad | Pre | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | |
| | Control | Pre | | | | | | | | | | |
| | | PIII(M4) | | | | | | | | | | |

Control =

Coad =

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

MIN/MAX = Minimum/Maximum

Pre = Day 0

PIII(M4) = Post Dose 3, Month 4

Template 23 Reverse Cumulative Distributions of Anti-CS Titres at Month 4, Coad and RTS,S groups (Per-Protocol Set)



RTS,S = Coad =

Template 24 Reverse Cumulative Distributions of Anti-Me titres at Month 4, Coad and Control groups (Per-Protocol Set)



Control = Coad =

200596 (MALARIA-073) Statistical Analysis Plan Final

# Template 25 Compliance to data capture per study group (Exposed Set)

| | | | ( | Coad/I | | grou<br>/Contr | | tal) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Do | ose 1 | Do | ose 2 | Do | se 3 | All | doses | Pe<br>subj | |
| Criteria | n | % | n | % | n | % | n | % | n | % |
| With visit done | | | | | | | | | | |
| With dose received | | | | | | | | | | |
| With Vitamin A received | | | | | | | | | | |
| With RTS,S AS01E dose received | | | | | | | | | | |
| With Measles and Rubella vaccine dose received | | | | | | | | | | |
| With Yellow fever dose received | | | | | | | | | | |
| With local solicited data available | | | | | | | | | | |
| With RTS,S AS01E local solicited data available | | | | | | | | | | |
| With Measles and Rubella local solicited data | | | | | | | | | | |
| available | | | | | | | | | | |
| With Yellow fever local solicited data available | | | | | | | | | | |
| With general solicited data available | | | | | | | | | | |

Coad =

RTS,S =

Control =

n = for each dose: number of subjects enrolled in the considered cohort and fulfilling specific criteria for the considered dose

for all doses: sum of n from individual doses

per subject : number of subjects enrolled in the considered cohort and fulfilling specific criteria for at least one dose % = percentage of doses with solicited/unsolicited data available among the number of administered doses

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 26 Incidence and nature of solicited and unsolicited symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | | An | y symp | tom | | | Genera | al sym | ptoms | ; | | Local | symp | toms | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | % CI | | | _ | | % CI | | | | | % CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | NA | NA | NA | NA | NA |
| Dose 2 | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | NA | NA | NA | NA | NA |
| Dose 3 | Coad | | | | | | | | | | | | | _ | | |
| (over 14 | RTS,S | | | | | | | | | | | | | | | |
| days) | | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | | | _ | | |
| - · | | - | | | _ | | - | | | | | 1 | | _ | | |
| Dose 3 | Coad | | | | | | _ | | | _ | | 1 | | + | | |
| (over 7 | RTS,S | | | _ | | | - | | | + | | | | | | |
| days) | Control | - | | _ | | | + | | - | + | | <u> </u> | | + | | |
| Overall/<br>dose | Coad | | | | | | | | | | | | | | | |
| dose | RTS,S | | | - | + | | + | | | + | | 1 | | | | |
| | Control | + | | + | + | | + | | + | + | | + | | + | | |
| | COITEO | | | + | | | + | | | + | | + | | | | |
| | | | | + | | | + | | | + | | | | 1 | | |
| Overall/ | Coad | 1 | | + | | | + | | 1 | + | | | | + | | |
| subject | Codd | | | | | | | | | | | | | | | |
| Cabject | RTS,S | | | + | | | + | | + | + | | | | + | + | |
| | Control | | | | | | + | | † | + | | 1 | | † | + | |
| | 30.1001 | | | + | | | + | | 1 | + | 1 | 1 | | t | + | |
| | | | | | | | + | | + | + | | 1 | | + | | |

Coad =

RTS,S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered For overall/dose:

N= number of administered doses

n%= number/percentage of doses followed by at least one type of symptom whatever the study vaccine administered 95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Over 14 days post vaccination at Dose 3

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 27 Incidence and nature of local solicited and unsolicited symptoms reported for each vaccine over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | | F | RTS,SAS0 | 1E | | | Meas | sles and F | Rubella | | | Y | ellow fev | er | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | - | 9 | 5% CI | | | | 9 | 5% CI | | | | 9 | 5% CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | Coad | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Dose 2 | Coad | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Dose 3 | Coad | | | | | | | | | | | | | | | |
| (over 14 days) | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |
| Dose 3 (over 7 | Coad | | | | | | | | | | | | | | | |
| days) | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |
| Overall/dose | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |
| Overall/subject | Coad | | | | | | | | | | | | | | | |
| • | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |

Coad =

RTS.S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

 $\label{eq:npercentage} \ \ n/\% = number/percentage \ of \ subjects \ presenting \ at \ least \ one \ type \ of \ symptom \ at \ the \ study \ vaccine \ site$ 

For overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom at the study vaccine site

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Over 14 days post vaccination at Dose 3

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

# Template 28 Incidence and nature of grade 3 solicited and unsolicited symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | | | Any s | ympton | 1 | | | General | symptom | <b>S</b> | | Lo | cal symp | toms | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 5% CI | | | | | 5% CI | | | | | % CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | NA | NA | NA | NA | NA |
| Dose 2 | Coad | | | | | | | | | | | | | | | T |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | NA | NA | NA | NA | NA |
| Dose 3 | Coad | | | | | | | | | | | | | | | |
| over 14 days) | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | | | | | |
| Overall/dose | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | | | | | |
| Overall/subject | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | | | | | |

Coad =

RTS.S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered For overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom whatever the study vaccine administered

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Over 14 days post vaccination at Dose 3

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 29 Incidence and nature of local grade 3 solicited and unsolicited symptoms reported for each vaccine over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | | | RTS,SAS | 01E | | | Mea | sles and | Rubella | | | | Yellow f | ever | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 9: | 5% CI | | | | 9 | 5% CI | | | | 9 | 5% CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | Coad | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Dose 2 | Coad | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Dose 3 | Coad | | | | | | | | | | | | | | | |
| (over 14 days) | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |
| Overall/dose | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |
| Overall/subject | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |

Coad =

RTS.S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects presenting at least one type of symptom at the study vaccine site For overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom at the study vaccine site

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Over 14 days post vaccination at Dose 3

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 30 Incidence and nature of solicited and unsolicited symptoms considered as causally related over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | | | Any sympt | om | | | Gen | eral symp | toms | | | Loc | al symptoi | ns | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 5% CI | | | | | 5% CI | | | | | % CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Dose 2 | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Dose 3 | Coad | | | | | | | | | | | | | | | |
| (over 14 days) | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | | | | | |
| Overall/dose | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | | | | | |
| Overall/subject | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | | | | | | | | | | |
| | Control | | | | | | | | | | | | | | | |

Coad =

RTS.S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered For overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom whatever the study vaccine administered

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Over 14 days post vaccination at Dose 3

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 31 Incidence and nature of solicited and unsolicited symptoms with considered causal relationship to vaccination, reported for each vaccine, over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | | F | RTS,SAS01 | E | | | Meas | les and R | Rubella | | | Ye | llow fev | er | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 9: | 5% CI | | | | 9 | 5% CI | | | | 95 | % CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | Coad | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Dose 2 | Coad | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Oose 3 | Coad | | | | | | | | | | | | | | | |
| over 14 days) | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |
| Overall/dose | Coad | | | | | | | | | | | | | | | |
| | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |
| )verall/subject | Coad | | | | | | | | | | | | | | | |
| • | RTS,S | | | | | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Control | NA | NA | NA | NA | NA | | | | | | | | | | |

Coad =

RTS.S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects presenting at least one type of symptom at the study vaccine site For overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom at the study vaccine site

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Over 14 days post vaccination at Dose 3

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 32 Incidence of solicited local symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | | | Coad | | | | | RTS,S | } | | | | Contro | l | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 9 | 5 % CI | | | | 9 | 5 % CI | | | | 9 | 5 % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | • | | • | | Dose 1 | • | ' | • | • | • | • | | • | |
| Pain | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Grade 3 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Redness (mm) | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Swelling (mm) | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | | | | - | | Dose 2 | | · | | | | | | | |
| Pain | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Grade 3 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Redness (mm) | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| , , | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Swelling (mm) | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | · | · | · | - | • | Dose 3 | | · | | | | | | | |
| Pain | All | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| Redness (mm) | All | | | | | | | | | | | | | | | |
| | >20.0 | | | | | | | | | | | | | | | |
| Swelling (mm) | All | | | | | | | | | | | | | | | |
| | >20.0 | | | | | | | | | | | | | | | |
| | <u> </u> | | | | - | Ov | erall/dos | е | • | | | | | | | |
| Pain | All | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| Redness (mm) | All | | | | | | | | | | | | | | | |
| | >20.0 | | | | | | | | | | | | | | | |
| Swelling (mm) | All | | | | | | | | | | | | | | | |
| | >20.0 | | | | | | | | | | | | | | | |

200596 (MALARIA-073) Statistical Analysis Plan Final

| | | | Coad | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Coad | | | | | RTS,S | | | | C | ontrol | | |
| | | | | | 95 9 | % CI | | | | 95 9 | % CI | | | | 95 9 | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | | | Overa | II/subject | | | | | | | | | |
| Pain | All | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| Redness (mm) | All | | | | | | | | | | | | | | | |
| | >20.0 | | | | | | | | | | | | | | | |
| Swelling (mm) | All | | | | | | | | | | | | | | | |
| | >20.0 | | | | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects reporting the symptom at least once

For Overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Solicited symptoms are reported over 14 days post Dose 3

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 33 Incidence of solicited local symptoms over 7 days post vaccination (Days 1-7) by dose and overall, by vaccine, per study group (Exposed Set)

| | | | | | Coad | | | | | RTS,S | | | | ( | Control | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI | | | | 95 | % CI | | | | 95 | % CI |
| Symptom | Product | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | | Dos | se 1 | | | | | | • | | • | _ | • | |
| Pain | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | Grade 3 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Redness (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Swelling (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | | • | • | Dos | se 2 | | ' | | ' | | | | | | • | |
| Pain | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | Grade 3 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Redness (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| Swelling (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | • | • | • | • | Dos | se 3 | | • | | ' | | | | | | • | |
| Pain | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | Grade 3 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | Grade 3 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | Grade 3 | | | | | | NA | NA | NA | NA | NA | | | | | |
| Redness (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| , , | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | $\top$ |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | 1 |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | $\top$ |

200596 (MALARIA-073) Statistical Analysis Plan Final

| | | | | Coad RTS,S 95 % CI 95 | | | | | | | | | | Stical A | Control | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI | | | ,. | | % CI | | | | 95 | % CI |
| Symptom | Product | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Swelling (mm) | RTSAS01E | All | | | | | | | | | 1 | | NA | NA | NA | NA | NA |
| 3( ) | | >20.0 | | | | | | | | | 1 | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | $\top$ |
| | | | | | Overa | II/dose | | | | | | | ' | | - | | |
| Pain | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | Grade 3 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | Grade 3 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | $\top$ |
| | | Grade 3 | | | | | | NA | NA | NA | NA | NA | | | | | |
| Redness (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| , , | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | 1 |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | |
| Swelling (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | • | • | • | Overall | /subjec | t | | | • | | • | • | • | • | · | |
| Pain | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | Grade 3 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | Grade 3 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | Grade 3 | | | | | | NA | NA | NA | NA | NA | | | | | |

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

| | | | | | Coad | | | | | RTS,S | | | | ( | Control | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI | | | - | 95 | % CI | | | | 95 9 | % CI |
| Symptom | Product | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Redness (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | |
| Swelling (mm) | RTSAS01E | All | | | | | | | | | | | NA | NA | NA | NA | NA |
| | | >20.0 | | | | | | | | | | | NA | NA | NA | NA | NA |
| | Measles and Rubella | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | |
| | Yellow fever | All | | | | | | NA | NA | NA | NA | NA | | | | | |
| | | >20.0 | | | | | | NA | NA | NA | NA | NA | | | | | $\top$ |

Coad =

RTS.S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects reporting the symptom at least once

For Overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Solicited symptoms are reported over 14 days post Dose 3

09-APR-2018 

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 34 Incidence of solicited general symptoms over 7 days post vaccination (Days 1-7) by dose and overall, per study group (Exposed Set)

| | | Coad 95 % CI | | | | | | | RTS | ,S | | | ( | ontro | ol | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95 | % CI | | | | 95<br>C | |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | U |
| | L | | | | Dos | e 1 | | | | 1 | | | | 1 | | _ |
| Drowsiness | All | | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Irritability / | All | | | | | | | | | | | | | | | |
| fussiness | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Loss of appetite | All | | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Temperature/ | All | | | | | | | | | | | | | | | |
| (Axillary) | Related | | | | | | | | | | | | | | | |
| (°C) | >39.0 | | | | | | | | | | | | | | | |
| | >39.0*Related | | | | | | | | | | | | | | | |
| Measles/rube | All | | | | | | | | | | | | | | | |
| lla-like rash | Related | | | | | | | | | | | | | | | |
| | >39.0 | | | | | | | | | | | | | | | |
| | >39.0*Related | | | | | | | | | | | | | | | |
| | | | | • | | | | | • | • | • | | ' | | • | |
| Drowsiness | All | | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Irritability / | All | | | | | | | | | | | | | | | |
| fussiness | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Loss of appetite | All | | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| | All | | | | | | | | | | | | | | | |
| (Axillary) | Related | | | | | | | | | | | | | | | |
| (°C) | >39.0 | | | | | | | | | | | | | | | |
| | >39.0*Related | | | | | | | | | | | | | | | |
| Measles/rube | | | | | | | | | | | | | | | | |
| lla-like rash | Related | | | | | | | | | | | | | | | |
| | >39.0 | | | | | | | | | | | L | | | | |
| | >39.0*Related | | | | | | | | | | | | | | | |

200596 (MALARIA-073) Statistical Analysis Plan Final

| | | Coad<br>95 % CI | | | | | | | RTS | ,S | | | ( | Contr | ol | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | % CI | | | | 95 | %<br>:I | |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | U<br>L |
| | | | | | Dos | se 3 | | | | | | | | | | |
| Drowsiness | All | | | | | | | | | | | | | | | ╙ |
| | Related | | | | | | | | | | | | | | | $\perp$ |
| | Grade 3 | | | | | | | $\perp$ | | | | | | | | $\perp$ |
| | Grade 3*Related | | | | | | | | | | | | | | | $\perp$ |
| Irritability / | All | | | | | | | $\perp$ | | | | | | | | $\perp$ |
| fussiness | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | $\perp$ |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Loss of appetite | All | | | | | | | | | | | | | | | |
| appente | Related | | | | | | | + | | + | 1 | | + | - | | + |
| | Grade 3 | | | | | | | | | | | | | | | $\top$ |
| | Grade 3*Related | | | | | | | | | | | | | | | $\top$ |
| Temperature/ | All | | | | | | | | | | | | | | | T |
| (Axillary) | Related | | | | | | | | | | | | | | | $\top$ |
| (°C) | >39.0 | | | | | | | | | | | | | | | $\top$ |
| , | >39.0*Related | | $\top$ | | | | | $\top$ | | | | | | | | $\top$ |
| Measles/rube | | | | | | | | | | | | | | | | + |
| lla-like rash | Related | | | | | | | | | | | | | | | + |
| | >39.0 | | 1 | | | | | 1 | | | | | | 1 | | $\top$ |
| | >39.0*Related | | 1 | | | | | 1 | | | | | | 1 | | $\top$ |
| | | | | 0 | veral | I/dose | 9 | • | | | | | | | - | |
| Drowsiness | All | | | | | T | | | | | | | | | | Т |
| | Related | | | | | | | | | | | | | | | $\top$ |
| | Grade 3 | | 1 | | | | | 1 | | | | | | 1 | | + |
| | Grade 3*Related | | | | | | | 1 | | | | | | | | + |
| Irritability / | All | | + | | | | | + | | | 1 | T | | + | | + |
| fussiness | Related | | 1 | | | 1 | | + | | | 1 | | | + | | $\top$ |
| | Grade 3 | | | | | | | | | | | | | | | $\top$ |
| | Grade 3*Related | | 1 | | | | | 1 | | | | | | 1 | | $\top$ |
| Loss of | All | | | | | | | | | | | | | | | $\top$ |
| appetite | | | _ | | | <u> </u> | | $\perp$ | | | | | $\perp$ | _ | | |
| | Related | | | | | _ | | | | | | _ | | _ | | $\bot$ |
| | Grade 3 | | _ | | <u> </u> | | | _ | | | | | | _ | | ┷ |
| | Grade 3*Related | | | | | _ | | _ | | | | | | | | $\perp$ |
| Temperature/ | | | 1 | | <u> </u> | 1 | 1 | $\bot$ | | | 1 | _ | 1 | _ | | 1 |
| (Axillary) | Related | | _ | | | ↓_ | | ┷ | | | _ | $oxed{oxed}$ | $\perp$ | _ | | 1 |
| (°C) | >39.0 | | _ | | <u> </u> | ↓ | | _ | | | 1 | _ | $\perp$ | | | $\perp$ |
| | >39.0*Related | | _ | | | 1 | _ | $\perp$ | | | 1 | $oxed{oxed}$ | $\perp$ | $\perp$ | | $\perp$ |
| Measles/rube | | | | | <u> </u> | | | $\perp$ | | | | $oxed{oxed}$ | $\perp$ | | | $\perp$ |
| lla-like rash | Related | | | | | | | | | | | | | | | |
| | >39.0 | | | | | | | | | | | | | | | |
| | >39.0*Related | | | | | | | | | | | | | | | |

200596 (MALARIA-073) Statistical Analysis Plan Final

| | | Coad 95 % CI | | | | | | | RTS | ,S | | | ( | Contr | ol | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95 | % CI | | | | 95<br>C | |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | U |
| | | | | Ov | erall | subje | ct | | | | | | | | | |
| Drowsiness | All | | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | T |
| Irritability / | All | | | | | | | | | | | | | | | |
| fussiness | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Loss of | All | | | | | | | | | | | | | | | |
| appetite | | | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | | | | | | |
| Temperature/ | All | | | | | | | | | | | | | | | |
| (Axillary) | Related | | | | | | | | | | | | | | | |
| (°C) | >39.0 | | | | | | | | | | | | | | | |
| | >39.0*Related | | | | | | | | | | | | | | | |
| Measles/rube | All | | | | | | | | | | | | | | | |
| -like rash | Related | $\top$ | + | | T | | | T | T | | | t | $\top$ | T | | $\top$ |
| | >39.0 | | | | | | | | | | | | $\top$ | 1 | | T |
| | >39.0*Related | | | 1 | | | | | | | | | | 1 | | Т |

Coad = RTS.S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects reporting the symptom at least once

For Overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Solicited symptoms are reported over 14 days post Dose 3

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 35 Maximum temperature reported during the 7-day (Days 1-7) post-vaccination period (overall doses), per study group (Exposed Set)

| | | | Co | ad N = | | | RT | S,S N = | | | Con | trol N : | = |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 959 | % CI | | | 95% | 6 CI | | | 95% | 6 CI |
| Characteristics | Categories | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Maximum | No fever | | | | | | | | | | | | |
| temperature | Unknown | | | | | | | | | | | | |
| | temperature | | | | | | | | | | | | |
| | [37.5-38.0] | | | | | | | | | | | | |
| | [38.1-38.5] | | | | | | | | | | | | |
| | [38.6-39.0] | | | | | | | | | | | | |
| | [39.1-39.5] | | | | | | | | | | | | |
| | [39.6-40.0] | | | | | | | | | | | | |
| | >40.0 | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

N = number of doses

n = number of doses in a given category

% = n / Number of doses with available results x 100

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Temperature is reported over 14 days post Dose 3

Template 36 Maximum temperature reported during the <7>-day (Days 1-<7>) post-vaccination period (<Dose 1>), per study group (Exposed Set)

| | | | Co | ad N = | 1 | | RT | S,S N = | | | Con | trol N = | = |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95 | % CI | | | 95% | 6 CI | | | 95% | 6 CI |
| Characteristics | Categories | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Maximum | No fever | | | | | | | | | | | | |
| temperature | [37.5-38.0] | | | | | | | | | | | | |
| | [38.1-38.5] | | | | | | | | | | | | |
| | [38.6-39.0] | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

N = number of subjects

n = number of subjects in a given category

% = n / Number of subjects with available results x 100

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 37 Percentage of subjects reporting unsolicited adverse events classified by MedDRA Primary System Organ Class and Preferred Term over 30 days (Days 1-30) post vaccination, per study group (Exposed Set)

| | | Coad N = 95% CI | | | | | RTS, | SN= | | | Contro | ol N = | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | 95% | 6 CI | | | 95% | CI |
| Primary System Organ | | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Class (CODE) | (CODE) | | | | | | | | | | | | |
| At least one symptom | | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting the symptom at least once

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Unsolicited adverse events are reported over 42 days post Dose 3

Template 38 Percentage of subjects reporting Serious Adverse Events (SAEs) classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post vaccination, per study group, Month 4.5 (Exposed Set)

| | | | | ad<br>= | | | | S,S<br>= | | | Con<br>N | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | | 95% | 6 CI | | | 95% | CI | |
| Primary System Organ<br>Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting the symptom at least once

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 39 Percentage of subjects with fatal SAEs classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post vaccination, per study group, Month 4.5 (Exposed Set)

| | | | Coa | d N = | | RTS,S N = | | | | | Contr | ol N = | • |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | 95% CI | | | | | 95% CI | | | |
| <b>Primary System Organ</b> | Preferred Term | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Class (CODE) | (CODE) | | | | | | | | | | | | |
| At least one symptom | | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting the symptom at least once

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 40 Percentage of subjects reporting SAEs with causal relationship to vaccination classified by MedDRA Primary System Organ Class and Preferred Term within 30 days post vaccination, per study group, Month 4.5 (Exposed Set)

| | | | Coa | d N = | | | RTS, | SN= | | Control N = | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | 95% CI | | | | | 95% CI | | |
| Primary System Organ | Preferred Term | | | | n | % | LL | UL | n | % | LL | UL |
| | (CODE) | | | | | | | | | | | |
| At least one symptom | | | | | | | | | | | | |

Coad =

RTS.S =

Control =

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of administered doses

n/% = number/percentage of doses with the symptom

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 41 Listing of SAEs reported until Month 4.5 visit, per study group (Exposed Set)

| Group | Sub. | Case | Age | Sex | Verbatim | Preferred | System | MA | Dose | Day | Duration | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | No. | ld | at | | | term | Organ | type | | of | | | |
| | | | onset | | | | Class | | | onset | | | |
| | | | (Year) | | | | | | | | | | |

Coad =

RTS,S =

Control =

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 42 Incidence of seizures by diagnostic certainty level within 7 days (1-7) post vaccination overall doses (Diagnostic certainty 1-5), per study group (Exposed Set)

| | | | Coad | N= | | | RTS,S | N: | | | Cont | rol N | = |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | Γ | | 95 | 5% | | | 95 | 5% CI |
| | | | | | | | | | ì | | | | |
| Characteristics | Categories | n | n/1000 | LL | UL | n | n/1000 | ᆸ | b | n | n/1000 | LL | UL |
| Generalized convulsive seizure | Level 1 to 3 | | | | | | | | | | | | |
| Convulsive seizure | Level 1 to 5 | | | | | | | | | | | | |
| Diagnostic certainty level | Level 1 | | | | | | | | | | | | |
| | Level 2 | | | | | Г | | | | | | | |
| | Level 3 | | | | | Γ | | | | | | | |
| | Level 4 | | | | | Г | | | | | | | |
| | Level 5 | | | | | Г | | | | | | | |

Coad =

RTS.S =

Control =

Total = Total

N = number of doses

n = number of doses in a given category

n/1000 = n / Number of doses with available results x 1000

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Level 1: Witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor

Level 2: History of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations

Level 3: History of unconsciousness AND other generalized motor manifestations

Level 4: Reported generalized convulsive seizure with insufficient evidence to meet the case definition

Level 5: Not a case of generalized convulsive seizure

Within 14 days post Dose 3

Template 43 Incidence of seizures by diagnostic certainty level and history of fever within 7 days (1-7) post vaccination overall doses (Diagnostic certainty 1-5), per study group (Exposed Set)

| | | | Coad | N= | | | RTS, | S N | = | | Conti | rol N | = |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 959 | 6 CI | | | 95 | % CI | | | 95 | % CI |
| Characteristics | Categories | n | n/1000 | LL | UL | n | n/1000 | LL | UL | n | n/1000 | LL | UL |
| Level 1 | History of fever | | | | | | | | | | | | |
| | No history of fever | | | | | | | | | | | | |
| Level 2 | History of fever | | | | | | | | | | | | |
| | No history of fever | | | | | | | | | | | | |
| Level 3 | History of fever | | | | | | | | | | | | |
| | No history of fever | | | | | | | | | | | | |
| Level 4 and 5 | History of fever | | | | | | | | | | | | |
| | No history of fever | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

Total = Total

N = number of generalized convulsive seizures

n = number of generalized convulsive seizures in a given category

% = n / Number of generalized convulsive seizures with available results x 100

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Level 1: Witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations

200596 (MALARIA-073) Statistical Analysis Plan Final

Level 2: History of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations

Level 3: History of unconsciousness AND other generalized motor manifestations

Level 4: Reported generalized convulsive seizure with insufficient evidence to meet the case definition

Level 5: Not a case of generalized convulsive seizure

Within 14 days post Dose 3

Template 44 Incidence of seizures by diagnostic certainty level and fever within 7 days (1-7) post vaccination overall doses (Diagnostic certainty 1-5), per study group (Exposed Set)

| | | | Coad | N = | : | | RTS, | S N | = | | Cont | rol N | = |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI<br>n n/1000 LL UL n n/1000 I | | | | % CI | | | 95 | % CI | | | |
| Characteristics | Categories | n | n/1000 | LL | UL | n | n/1000 | LL | UL | n | n/1000 | LL | UL |
| Level 1 | <38°C | | | | | | | | | | | | |
| | ≥38°C | | | | | | | | | | | | |
| | Missing temperature | | | | | Г | | | | Г | | | |
| Level 2 | <38°C | | | | | Г | | | | Г | | | |
| | ≥38°C | | | | | | | | | | | | |
| | Missing temperature | | | | | | | | | | | | |
| Level 3 | <38°C | | | | | | | | | | | | |
| | ≥38°C | | | | | | | | | | | | |
| | Missing temperature | | | | | | | | | | | | |
| Level 4 and 5 | <38°C | | | | | | | | | | | | |
| | ≥38°C | | | | | | | | | | | | |
| | Missing temperature | | | | | | | | , i | | | | |

Coad =

RTS,S =

Control =

Total = Total

N = number of generalized convulsive seizures

n = number of generalized convulsive seizures in a given category

% = n / Number of generalized convulsive seizures with available results x 100

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Level 1: Witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations

Level 2: History of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations

Level 3: History of unconsciousness AND other generalized motor manifestations

Level 4: Reported generalized convulsive seizure with insufficient evidence to meet the case definition

Level 5: Not a case of generalized convulsive seizure

Within 14 days post Dose 3

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 45 Incidence of concomitant medication administered during the <30day (Days 1-30)> post-vaccination period by dose and overall, per study group (Exposed Set)

| | | Coad 95% CI | | | | | RTS,S | ; | | | С | ontro | ol | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 95 | % CI | | | | 95 | % CI | | | | 95 | % CI |
| | N | | | | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | D | ose 1 | | | | | | | | | |
| Any antipyretic | | | | | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | | | | | |
| | | | | D | ose 2 | | | | | | | | | |
| Any antipyretic | | | | | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | | | | | |
| | | | | D | ose 3 | | | | | | | | | |
| Any antipyretic | | | | | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | | | | | |
| | | | | Ove | rall/do | se | | | | | | | | |
| Any antipyretic | | | | | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | | | | | |
| | | | | Overa | ıll/sub | ject | | | | | | | | |
| Any antipyretic | | | | | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | | | | | |

Coad =

RTS,S =

Control =

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects who started to take the specified concomitant medication at least once during the mentioned period

For overall/dose:

N= number of administered doses

During the < 42-day> post-vaccination period post Dose 3

Template 46 Number (%) of subjects with serious adverse events including number of events reported during the study period (Exposed Set)

| | | | | Coad | N = | F | RTS,S | N = | С | Control N = | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System<br>Organ Class | Preferred Term<br>(CODE) | n* | n | % | n* | n | % | n* | n | % |
| SAE | At least one symptom | | | | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | | | | |
| Related SAE | At least one symptom | | | | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | | | | |
| Fatal SAE | At least one symptom | | | | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | | | | |
| Related fatal<br>SAE | At least one symptom | | | | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | | | | |

Coad =

RTS,S =

Control =

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

200596 (MALARIA-073) Statistical Analysis Plan Final

Template 47 Solicited and unsolicited symptoms, classified by MedDRA Primary System Organ Class and Preferred Term within the 42-day (Days 1-42) post-vaccination period including number of events - SAE excluded (Exposed Set)

| | | C | CoadN = | | | S,S N | = | Control N = | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Primary System<br>Organ Class<br>(CODE) | Preferred Term<br>(CODE) | n* | n | % | n* | n | % | n* | n | % |
| At least one symptom | | | | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | | | | |

Coad =

RTS,S =

Control =

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

Template 48 Listing of dropouts due to AEs, SAEs and solicited symptoms (Exposed Set)

| Group | Study -<br>Subject | Country | Gender | 1 | AE<br>Descripti<br>on | SAE | Causality | Type of discontinuati on |
|---|---|---|---|---|---|---|---|---|